CLINICAL TRIAL: NCT03087071
Title: A Phase II Enrichment Study of Panitumumab as a Single Agent or in Combination With Trametinib in Anti-EGFR-Refractory Stage IV Colorectal Cancer Patients
Brief Title: Panitumumab With or Without Trametinib in Treating Patients With Stage IV Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0338; NCI-2017-00868 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0338 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: EGFR NP_005219.2:p.S492R; KRAS Gene Mutation; MAP2K1 Gene Mutation; Metastatic Colorectal Adenocarcinoma; Refractory Colorectal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (panitumumab) (Experimental): Patients with EGFR ectodomain mutation receive panitumumab IV over 30-90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Cohort 2.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Panitumumab
- Cohort 2 (panitumumab, trametinib) (Experimental): Patients with KRAS, NRAS, or BRAF mutation receive trametinib PO QD on days 1-14 and panitumumab as in Cohort 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Panitumumab; Drug: Trametinib
- Cohort 3 (panitumumab) (Experimental): Patients without EGFR ectodomain, KRAS, NRAS, or BRAF mutation receive panitumumab as in Cohort 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Cohort 2.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Panitumumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
  Arms: Cohort 2 (panitumumab, trametinib)

SUMMARY:
This phase II clinical trial studies how well panitumumab with or without trametinib works in treating patients with stage IV colorectal cancer. Immunotherapy with monoclonal antibodies, such as panitumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving panitumumab with or without trametinib may work better in treating patients with stage IV colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor efficacy of panitumumab monotherapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently have detectable EGFR ectodomain mutation post-progression in circulating free tumor deoxyribonucleic acid (DNA).

II. To evaluate the anti-tumor efficacy of panitumumab and trametinib combination therapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently have detectable levels of KRAS, NRAS, and/or BRAF mutation post-progression in circulating free tumor DNA.

III. To evaluate the anti-tumor efficacy of panitumumab monotherapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently do not have detectable KRAS, NRAS, BRAF, or EGFR ectodomain mutation post-progression in circulating free tumor DNA.

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of panitumumab and trametinib combination therapy.

II. To evaluate the anti-tumor efficacy of panitumumab and trametinib combination therapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who progressed on prior anti-EGFR therapy, developed detectable EGFR ectodomain mutations, and progress through retreatment with panitumumab.

III. To evaluate the anti-tumor efficacy of panitumumab and trametinib combination therapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who progressed on prior anti-EGFR therapy, did not develop detectable mutations in KRAS, NRAS, BRAF, or EGFR ectodomain, and progress through retreatment with panitumumab.

IV. To evaluate clinical outcomes with panitumumab monotherapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently have detectable EGFR ectodomain mutation post-progression in circulating free tumor DNA.

V. To evaluate clinical outcomes with panitumumab and trametinib combination therapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently have detectable levels of KRAS, NRAS, and/or BRAF mutation post-progression in circulating free tumor DNA.

VI. To evaluate clinical outcomes with panitumumab monotherapy in patients who were initially KRAS/NRAS/BRAF wild-type at baseline who have progressed on prior anti-EGFR therapy and subsequently do not have detectable KRAS, NRAS, BRAF, or EGFR ectodomain mutation post-progression in circulating free tumor DNA.

VII. To study the biological basis of development of primary and secondary resistance to anti-EGFR antibodies and MEK inhibitors.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: Patients with EGFR ectodomain mutation receive panitumumab intravenously (IV) over 30-90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Cohort 2.

COHORT 2: Patients with KRAS, NRAS, or BRAF mutation receive trametinib orally (PO) once daily (QD) on days 1-14 and panitumumab as in Cohort 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

COHORT 3: Patients without EGFR ectodomain, KRAS, NRAS, or BRAF mutation receive panitumumab as in Cohort 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Cohort 2.

After completion of study treatment, patients are followed up for 4 weeks and then every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal adenocarcinoma, with metastatic disease documented on diagnostic imaging studies
* Progression during or within 6 months after fluoropyrimidine, irinotecan, and oxaliplatin; for oxaliplatin-based therapy, failure of therapy will also include patients who progressed within 12 months of adjuvant therapy and patients who had oxaliplatin discontinued secondary to toxicity or allergic reaction; patients with a known history of Gilbert's disease who cannot receive irinotecan or patients who are intolerant of irinotecan or fluoropyrimidine are eligible
* Confirmed wild-type status in KRAS exons 2, 3, and 4; NRAS exons 2, 3, and 4; and BRAF, by standard of care testing of tumor specimen; tissue used for testing may have been collected prior to treatment with anti-EGFR therapy
* Patient must have been already tested and have available results of the mutations status of KRAS/NRAS/BRAF/MEK (MAP2K1) and EGFR from the circulating tumor DNA within 10 weeks prior to starting study therapy
* Previous treatment with anti-EGFR therapy with evidence of clinical benefit, as defined by complete response, partial response, or prolonged stable disease with 16 or more weeks of treatment without radiographic progression, as assessed by the treating physician and documented in the medical record; this treatment may have occurred at any point in the patient's clinical course for treatment of metastatic colorectal cancer
* Ultimate progression through previous treatment with anti-EGFR therapy, with documented clinical progression; patients who discontinued anti-EGFR therapy for any other reason, such as decline in performance status, hypersensitivity, or other adverse effects of therapy, are not eligible
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0) =< grade 1 (except =< grade 2 for alopecia peripheral neuropathy)
* Radiographically measurable disease present per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Blood counts performed within 3 weeks prior to starting study therapy must have absolute neutrophil count >= 1,500/mm^3
* Blood counts performed within 3 weeks prior to starting study therapy must have platelets >= 100,000/mm^3
* Blood counts performed within 3 weeks prior to starting study therapy must have hemoglobin >= 9 g/dL
* Liver function tests performed within 3 weeks prior to starting study therapy must have total bilirubin =< 1.5 x upper limit of normal (ULN)
* Liver function tests performed within 3 weeks prior to starting study therapy must have alanine aminotransferase and aspartate aminotransferase =< 2.5 x ULN (or =< 5 x ULN if liver metastases are present)
* Liver function tests performed within 3 weeks prior to starting study therapy must have albumin >= 2.5 g/dL
* Serum creatinine performed within 3 weeks prior to starting study therapy must be =< 1.5 x ULN, or have calculated creatinine clearance (using Cockcroft-Gault formula) of >= 50 mL/minute
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) performed within 3 weeks prior to starting study therapy must be =< 1.5 x ULN
* Left ventricular ejection fraction (LVEF) >= lower limit of normal (LLN) by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 3 weeks prior to starting study therapy
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization and must agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment
* Ability to sign informed consent form; informed consent form for this study must be signed prior to the performance of any study-specific procedures and initiation of any study therapy
* Ability to swallow and retain oral medication, with no clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* In cohort 1, must have EGFR S492R or other ectodomain mutation detected from circulating tumor DNA from plasma collected after progression on prior anti-EGFR therapy; may have a concomitant mutation in KRAS, NRAS, or BRAF, if there is at least a 5-fold higher allele frequency of the most prevalent EGFR mutation than the most prevalent KRAS/NRAS/BRAF mutation
* In cohort 2, must have one or more mutations found in KRAS exon 2, 3, or 4; NRAS exon 2, 3, or 4; BRAF codon 600; or in MEK (MAP2K1); may have a concomitant EGFR ectodomain mutation, if the most prevalent EGFR ectodomain mutation does not have over a 5-fold higher allele frequency than the most prevalent KRAS/NRAS/BRAF mutation
* In cohort 3, must not have EGFR ectodomain mutation or any mutations in KRAS, NRAS, or BRAF

Exclusion Criteria:

* Past treatment with any MEK or ERK inhibitor
* Previous retreatment with anti-EGFR therapy following progression on initial course of anti-EGFR therapy
* Known untreated brain metastasis or brain metastasis treated within 3 months prior to enrollment in this trial
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* History of interstitial lung disease or pneumonitis
* History of any other malignancy within 3 years, except for adequately treated carcinoma in situ of the cervix or non-melanoma skin cancer and/or subjects with indolent second malignancies are eligible
* Prior treatment within 21 days of the first dose of study drug with any other chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment, or failure to recover from adverse effects of prior therapies administered over 4 weeks prior to study day 1; all toxicities from prior therapies must be =< grade 1 (or =< grade 2 for alopecia or peripheral neuropathy); prior systemic treatment in the adjuvant setting is allowed
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomization and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to randomization
* Impaired cardiac function or clinically significant cardiac disease, as defined: a) left ventricular ejection fraction < lower limit of normal (LLN) on multiple gated acquisition scan (MUGA) or echocardiogram; b) congenital long QT syndrome or family history of unexpected sudden cardiac death; c) corrected QT (QTc) corrected with Bazett's formula (QTcB) >= 480 ms.; d) history or evidence of current clinically significant uncontrolled arrhythmias; note subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible; e) history of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization; f) history or evidence of current >= class II congestive heart failure as defined by New York Heart Association (NYHA); g) treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy; h) patients with intra-cardiac defibrillators
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent, or compliance to the study procedures
* History of retinal vein occlusion (RVO)
* Pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment
* History of organ allograft or other history of immunodeficiency
* Inability or unwillingness to comply with study and/or follow-up requirements
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO)
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection; subjects with laboratory evidence of cleared HBV and HCV infection will be permitted
* Current use of a prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 24 months
  Will be evaluated along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Complete response | Up to 24 months
  The incidence rates will be estimated, along with the exact 95% confidence intervals.
Partial response | Up to 24 months
  The incidence rates will be estimated, along with the exact 95% confidence intervals.
Stable disease | Up to 24 months
  The incidence rates will be estimated, along with the exact 95% confidence intervals.
Progression-free survival (PFS) | Up to 24 months
  The probability of PFS will be estimated using the method of Kaplan and Meier. The two-sided log-rank test will be used to assess the differences between groups.
Overall survival (OS) | Up to 24 months
  The probability of OS will be estimated using the method of Kaplan and Meier. The two-sided log-rank test will be used to assess the differences between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Parseghian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org